CLINICAL TRIAL: NCT05287867
Title: A Trial of Platelet Injections for Treatment of Painful Degenerative Disc Disease
Brief Title: Trial for Treating Painful Degenerative Disc Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Regenexx, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: RGX2021-01
Record Dates: First submitted 2022-03-04; First posted 2022-03-18 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Platelet treatment (Experimental): A series of two treatments spaced 4 weeks apart that include platelet-rich plasma (PRP). platelet lysate (PL), and platelet poor plasma (PPP).
  Interventions: Biological: Platelet-rich plasma (PRP), Platelet lysate (PL), and Platelet Poor Plasma (PPP)
- Sham procedure (Sham Comparator): A series of two sham procedures spaced 4 weeks apart.
  Interventions: Other: Sham procedure

INTERVENTIONS:
Biological: Platelet-rich plasma (PRP), Platelet lysate (PL), and Platelet Poor Plasma (PPP) — Approx 161-420cc autologous blood is drawn and processed into PPP, PRP, and PL, amount dependent on condition. Using sterile technique with patient sedated, US or x-ray is used to guide needles bilaterally into multifidus, specifically LM, TF, IAF. Once the lamina is reached the physician injects 2.5 cc of PPP into the multifidus muscle on one side and then repeat this on the opposite side for each level. The physician guides a needle into the supraneural transforaminal space to perform an epidural injection with 2cc of 4x PL and 1 cc of 0.5% ropivacaine. Next, a needle will then be guided into the facet joint to perform an intra-articular injection with 1cc of 14x PRP. Any tendon insertion areas will be injected using ultrasound guidance with platelet lysate dextrose. The supraspinous/interspinous, SI ligaments at the involved degenerative levels will be injected with 4x PL/12.5% dextrose/0.125% ropivacaine. If L5/S1 is involved, the iliolumbar ligaments will also be injected.
  Arms: Platelet treatment
Other: Sham procedure — Approximately 161-420 cc of autologous blood is drawn to maintain patient blinding. While lying prone, the patient's back will be exposed and prepped sterilely.
  Provider puts patient in conscious sedation and several needles are placed into the low back. The provider inserts needle into the facet joint and then removes. Then inserts the needle midline to ligament and removes (1 needle per level) mimicking normal needle placement, but not injecting anything.
  Arms: Sham procedure

SUMMARY:
To evaluate and compare two platelet-based treatments of the functional spinal unit spaced 4 weeks apart to sham procedures for the treatment of degenerative disc disease.

DETAILED DESCRIPTION:
This is a single-blind, randomized, placebo-controlled study using platelet-based treatment to the functional spinal unit .in a series of 2 treatments 4 weeks apart to treat painful lumbar degenerative disc disease. Randomization is 2:1, with 28 in the treatment group and 14 in the sham control group.

A pretreatment visit will occur at or before the time of enrollment; follow-up visits will occur at the clinical site at 3- and 12 months post injection. Target enrollment is 42 subjects. Patients in the control group can crossover to the treatment group after 3-month follow-up. Crossover patients then follow the treatment group follow-up timeline based on their second real treatment. Subjects will complete the study following the 1-year follow-up visit.

The primary objective of this study is to observe the improvement in subject-reported clinical outcomes from baseline to 3 months after 2nd treatment and between groups at 3 months, with continued evaluation of efficacy and durability up to 12 months. Questionnaires are completed at 1, 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary signature of the IRB approved Informed Consent,
* Skeletally mature Male or Female ages 25 to 65
* Maximum of 3 levels degenerative disc disease without significant spondylolisthesis in the area c/w the pain (grade 1 with less than or equal to 10% vertebral body)
* Chronic back and/or leg pain having failed conservative treatment (e.g. NSAIDs, physician initiated physical therapy) for at least 6 months
* MRI and physical examination consistent with painful Degenerative Disc Disease
* Failure of epidural steroid injection, facet injection, medial branch block, radiofrequency ablation or physical therapy
* Instability as seen on MRI, flexion-extension x-ray, or physical deformity as seen on MRI c/w degenerative instability (facet hypertrophy, loss of disc height, spondylolisthesis, laterolisthesis, osteophytes)
* A lumbar surgery candidate (will need to specify which surgery, ie. fusion, decompression, etc)
* Is independent, ambulatory, and can comply with all post-operative evaluations and visits

Exclusion criteria:

* Evidence of more than moderate central canal or foraminal stenosis
* Smoker or cessation for less than 6 weeks
* Untreated underlying psychological conditions (e.g. depression, chronic pain syndrome, etc.) as a contributor to chronic pain
* Prior epidural steroid injection within the past 8 weeks
* Degenerative scoliosis if cob angle over 10 degrees
* Undergone previous Regenexx lumbar procedure
* Standing intolerance (patient cannot stand longer than 30 minutes)
* Inflammatory or auto-immune based pathology (e.g., rheumatoid arthritis, systemic lupus erythematosus, psoriatic arthritis, polymyalgia, polymyositis, gout pseudogout)
* Severe neurogenic inflammation of the cutaneous nerves
* Condition represents a worker's compensation case
* Currently involved in a health-related litigation procedure
* Is pregnant
* Bleeding disorders
* Currently taking anticoagulant or immunosuppressive medication
* Allergy or intolerance to study medication
* Use of chronic opioid
* Documented history of drug abuse within six months of treatment
* Central sensitization
* Hypermobile or EDS
* 19) Any other condition, that in the opinion of the investigator, that would preclude the patient from enrollment

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-05-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Scale (NPS) | 3-months after 2nd treatment
  Difference in Numeric Pain Scale group differences (scale 0-10, where 0=no pain and 10=worst possible pain
Modified Single Assessment Numerical Evaluation (SANE) scores | 3-months after 2nd treatment
  Difference in modified Single Assessment Numerical Evaluation score group differences; scores range from 0-100 where 0=no improvement and 100=100% improved

SECONDARY OUTCOMES:
Mean modified SANE scores | 1-month, 3-months, 6 months, 12 months
  Average SANE scores post-treatment; scores range from 0-100 where 0=no improvement and 100=100% improved
Numeric Pain Scale (NPS) | Baseline, 1-month, 3-months, 6 months, 12 months
  Changes in NPS from pre to post treatment; scale ranges from 0-10 where 0=no pain and 10=worst possible pain
Functional Rating Index (FRI) | Baseline, 1-month, 3-months, 6 months, 12 months
  Changes in FRI from pre to post treatment and between group differences at 1 and 3 months; scales 0-100% where 0%=no disability and 100%=very severe disability
Oswestry Disability Index (ODI) | Baseline, 1-month, 3-months, 6 months, 12 months
  Changes in ODI from pre to post and between group differences at 1 and 3 months; scales 0-100% where 0%=no disability and 100%=very disabled.
Incidence rate of adverse events | 1 month, 3 months, 6 months and 12 months
  Incidence of adverse events after treatment
Incidence rate of surgical/other treatment interventions | 1 month, 3 months , 6 months and 12 months
  Incidence of surgical/other treatment interventions after treatment
Pain medications | 1 month, 3 months, 6 months and 12 months
  Changes in medications from pre to post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Centeno, MD, Principal Investigator — Centeno-Schultz Clinic
Locations (2):
- United States (2):
  - Centeno-Schultz Clinic, Broomfield, Colorado
  - Centeno-Schultz Clinic, Lone Tree, Colorado

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Manchikanti L, Singh V, Falco FJ, Cash KA, Pampati V. Evaluation of the effectiveness of lumbar interlaminar epidural injections in managing chronic pain of lumbar disc herniation or radiculitis: a randomized, double-blind, controlled trial. Pain Physician. 2010 Jul-Aug;13(4):343-55. PMID 20648203
- [Background] Ravindra VM, Senglaub SS, Rattani A, Dewan MC, Hartl R, Bisson E, Park KB, Shrime MG. Degenerative Lumbar Spine Disease: Estimating Global Incidence and Worldwide Volume. Global Spine J. 2018 Dec;8(8):784-794. doi: 10.1177/2192568218770769. Epub 2018 Apr 24. PMID 30560029
- [Background] Rodrigues SV, Acharya AB, Thakur SL. Platelet-rich plasma. A review. N Y State Dent J. 2012 Jan;78(1):26-30. PMID 22474794
- [Background] Capelli C, Domenghini M, Borleri G, Bellavita P, Poma R, Carobbio A, Mico C, Rambaldi A, Golay J, Introna M. Human platelet lysate allows expansion and clinical grade production of mesenchymal stromal cells from small samples of bone marrow aspirates or marrow filter washouts. Bone Marrow Transplant. 2007 Oct;40(8):785-91. doi: 10.1038/sj.bmt.1705798. Epub 2007 Aug 6. PMID 17680021
- [Background] Centeno CJ, Schultz JR, Cheever M, Freeman M, Faulkner S, Robinson B, Hanson R. Safety and complications reporting update on the re-implantation of culture-expanded mesenchymal stem cells using autologous platelet lysate technique. Curr Stem Cell Res Ther. 2011 Dec;6(4):368-78. doi: 10.2174/157488811797904371. PMID 22023622
- [Background] Centeno C, Markle J, Dodson E, Stemper I, Hyzy M, Williams C, Freeman M. The use of lumbar epidural injection of platelet lysate for treatment of radicular pain. J Exp Orthop. 2017 Nov 25;4(1):38. doi: 10.1186/s40634-017-0113-5. PMID 29177632
- [Background] Williams C, Jerome M, Fausel C, Dodson E, Stemper I, Centeno C. Regenerative Injection Treatments Utilizing Platelet Products and Prolotherapy for Cervical Spine Pain: A Functional Spinal Unit Approach. Cureus. 2021 Oct 8;13(10):e18608. doi: 10.7759/cureus.18608. eCollection 2021 Oct. PMID 34659923
- [Background] Phillips FM, Slosar PJ, Youssef JA, Andersson G, Papatheofanis F. Lumbar spine fusion for chronic low back pain due to degenerative disc disease: a systematic review. Spine (Phila Pa 1976). 2013 Apr 1;38(7):E409-22. doi: 10.1097/BRS.0b013e3182877f11. PMID 23334400